CLINICAL TRIAL: NCT00001409
Title: A Phase I/II Pilot Study of the Safety of the Adoptive Transfer of Syngeneic Gene-Modified Cytotoxic T Lymphocytes in HIV Infected Identical Twins
Brief Title: Genetically Modified Lymphocytes to Treat HIV-Infected Identical Twins - Study Modifications
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940206; 94-I-0206
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-06

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infection
Keywords: AIDS; Gene Therapy; T Cell Universal Receptor; Ex Vivo Activation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2

SUMMARY:
Certain patients enrolled in NIH protocol 94-I-0206 at the Clinical Center may be eligible to participate in one or more of the following new options:

* Donor/recipient extension phase - Both the recipient (HIV-infected twin) and donor (non-infected twin) will participate in this extension of the CD4-zeta gene therapy study. It will evaluate the safety and activity of infusing gene-modified CD4+ cells as well as the modified CD8+ cells.
* Corticosteroid administration - A corticosteroid, such as prednisone, hydrocortisone or prednisolone, will be added to the interleukin-2 (IL-2) regimen for preventing or treating side effects of IL-2 such as fever and other flu-like symptoms.
* Extended follow-up - A more intensive follow-up will be scheduled for patients with substantial numbers of lymphocytes that harbor the CD4-zeta gene. Every 3 months, participants will have blood tests and specialized tests of CD4 counts, HIV-1 viral load and numbers of circulating cells containing the CD4-zeta gene every 3 months> the frequency of follow-up visits may be reduced as time goes by.
* IL-2 continuation - Participants will continue to receive periodic treatment with IL-2 to see how long the genetically modified cells persist in the bloodstream and to evaluate the long-term response to IL-2.
* Home treatment with interleukin-2 - Participants may receive future IL-2 treatment cycles at home. Home treatment involves less frequent data and safety monitoring and no medical evaluations at the Clinical Center except at the beginning of each cycle.

DETAILED DESCRIPTION:
Open-label, comparative, sequentially randomized treatment with genetically unmodified or modified ex vivo-expanded T-lymphocytes in patients with HIV infection who possess a seronegative syngeneic twin. Genetic modification consists of introduction of a gene for HLA-unrestricted "universal" receptors specific for the gp120 HIV envelope protein. Treatment is divided into Periods I and II.

ELIGIBILITY:
INCLUSION CRITERIA:

An identical twin pair, one of whom is seropositive for HIV, the other twin seronegative, by standard ELISA, PCR, and Western blot testing.

Patients whose CD4+ count is less than 500/mm(3) at entry must have been on FDA-approved or expanded-access antiretroviral agent(s) for at least 2 months.

Patients with Kaposi's sarcoma are eligible for this study, but must not have received any systemic therapy for KS within 4 weeks prior to entry. The diagnosis of KS must have been confirmed by biopsy.

Anticipated survival greater than 6 months and Karnofsky Performance Status greater than or equal to 60%.

Males or females 18 years of age or older. Every effort will be made to include both genders.

Free from serious psychological or emotional illness and able to provide written informed consent.

EXCLUSION CRITERIA - RECIPIENT:

Lymphoma.

Unwillingness to comply with current NIH Clinical Center guidelines concerning appropriate notification of all current sexual partners of an individual regarding his or her HIV positive sero-status and the risk of transmission of HIV infection.

Recent history of substance abuse unless evidence is provided of an ongoing therapeutic intervention (i.e. medical therapy or counseling) to control such abuse.

Pregnancy at entry or unwillingness to practice barrier birth control or abstinence during the study.

EXCLUSION CRITERIA - DONOR:

Untreated or inadequately treated medical condition (e.g., cardiopulmonary disease, acute infection) which, in the judgement of the Principal Investigator, precludes apheresis.

Serologic positivity for Epstein Barr virus, Cytomegalovirus, Hepatitis B or Hepatitis C if and only if the recipient twin tests seronegative for the corresponding virus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1994-09; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lane HC, Zunich KM, Wilson W, Cefali F, Easter M, Kovacs JA, Masur H, Leitman SF, Klein HG, Steis RG, et al. Syngeneic bone marrow transplantation and adoptive transfer of peripheral blood lymphocytes combined with zidovudine in human immunodeficiency virus (HIV) infection. Ann Intern Med. 1990 Oct 1;113(7):512-9. doi: 10.7326/0003-4819-113-7-512. PMID 1975487
- [Background] Koenig S, Conley AJ, Brewah YA, Jones GM, Leath S, Boots LJ, Davey V, Pantaleo G, Demarest JF, Carter C, et al. Transfer of HIV-1-specific cytotoxic T lymphocytes to an AIDS patient leads to selection for mutant HIV variants and subsequent disease progression. Nat Med. 1995 Apr;1(4):330-6. doi: 10.1038/nm0495-330. PMID 7585062
- [Background] Roberts MR, Qin L, Zhang D, Smith DH, Tran AC, Dull TJ, Groopman JE, Capon DJ, Byrn RA, Finer MH. Targeting of human immunodeficiency virus-infected cells by CD8+ T lymphocytes armed with universal T-cell receptors. Blood. 1994 Nov 1;84(9):2878-89. PMID 7949163